CLINICAL TRIAL: NCT05903963
Title: Evaluation of Renal Protection Of Dexmedetomidine Versus Midazolam As a Sedative For Septic Patients In Intensive Care Unit
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Marlin Zarif Shehata Yousef, Ass. lecturer of anesthesia and pain medicine, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 335-2022
Record Dates: First submitted 2023-05-30; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Renal Failure
MeSH Terms: conditions — Renal Insufficiency | interventions — Midazolam; Dexmedetomidine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Midazolam group (Active Comparator)
  Interventions: Drug: Midazolam
- dexmedetomidine group (Active Comparator)
  Interventions: Drug: dexmedetomidine

INTERVENTIONS:
Drug: Midazolam — midazolam infusion by 0.03-0.3mg/kg in increments of 1-2.5mg followed by Maintenance dose: 0.03-0.2mg/kg/hour for midazolam.
  Arms: Midazolam group
Drug: dexmedetomidine — dexmedetomidine infusion 1 µg/kg dexmedetomidine for 10 minutes followed by a continuous IV infusion at 0.2-0.3 µg/kg/hour .
  Arms: dexmedetomidine group

SUMMARY:
Evaluation of Renal Protection Of Dexmedetomidine Versus Midazolam As a Sedative For Septic Patients In Intensive Care Unit

ELIGIBILITY:
Inclusion Criteria:

* Age (18-80) years old. sex:both male and female.
* intubated and mechanically ventilated patients.

Exclusion Criteria:

* 1.Patient's relatives refusal. 2. burns as admitting diagnoses. 3.patients with any renal pathology(such as chronic glomerulonephritis, pyelonephritis and diabetic nephropathy).

  4. pregnancy or lactation. 5. serious central nervous system pathology (acute stroke, uncontrolled seizures, severe dementia).

  6. acute hepatitis or severe liver disease (Child-Pugh class C). 7. unstable angina or acute myocardial infarction, left ventricular ejection fraction less than 30%, heart rate less than 50/min, second- or third-degree heart block, or systolic blood pressure less than 90 mm Hg despite continuous infusions of 2 vasopressors before the start of study drug infusion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05-22 (Actual); Primary Completion 2023-11-12 (Estimated); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute kidney injury | 5 days
  urinary kidney injury molecule

SECONDARY OUTCOMES:
length of ICU stay | 10 days
  days of ICU stay

CONTACTS AND LOCATIONS:
Locations (1):
- Marlin Zarif Shehata, Minya, Egypt